CLINICAL TRIAL: NCT05862181
Title: Efficacy and Safety of HepaSphere Drug-eluting Bead Transarterial Chemoembolization Combined With Hepatic Arterial Infusion Chemotherapy in Advanced Hepatocellular Carcinoma
Brief Title: The Comparison Between HepaSphere Drug-eluting Bead Transarterial Chemoembolization Combined With Hepatic Arterial Infusion Chemotherapy in Advanced Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Other Study IDs: HCC-HEPA-HAIC-001
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-03

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
Keywords: HepaSphere; Transarterial chemoembolization; TACE; Hepatic Arterial Infusion Chemotherapy; HAIC

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HEPA-HAIC group: HEPA-HAIC group is composed of advanced HCC patients treated with HepaSphere DEB-TACE combined with HAIC as the interventional therapy
  Interventions: Procedure: DEB-TACE plus HAIC or HAIC alone
- HAIC group: HAIC group is composed of advanced HCC patients treated with only HAIC as the interventional therapy
  Interventions: Procedure: DEB-TACE plus HAIC or HAIC alone

INTERVENTIONS:
Procedure: DEB-TACE plus HAIC or HAIC alone — the patients received DEB-TACE plus HAIC or HAIC at least twice during this observational study

SUMMARY:
Transarterial chemoembolization (TACE) is widely applied and shows good efficacy in advanced hepatocellular carcinoma (HCC). Recently, hepatic arterial infusion chemotherapy (HAIC) has also gained popularity in the treatment of HCC. Several studies have described the comparison between HAIC and TACE or TACE combined with HAIC. However, the evaluation between TACE plus HAIC and HAIC is rarely reported. Here, we will evaluate the performance of HepaSphere DEB-TACE combined with HAIC (HEPA-HAIC) comparing to HAIC in patients with advanced HCC

DETAILED DESCRIPTION:
This is a double-arm, retrospective, observational study. The patients diagnosed as advanced HCC and treated with HepaSphere plus HAIC or single HAIC in the interventional therapy department of Peking University Cancer Hospital & Institute from May 2018 to May 2022. These patients are grouped into two cohorts. One is HEPA-HAIC group, the other is HAIC group. To access the effect of HepaSphere plus HAIC and single HAIC on the treatment of advanced HCC, the treatment efficacy and safety will be analyzed between these two cohorts. To avoid the selection bias, Propensity score matching (PSM) will be also conducted. The primary endpoints are progression-free survival (PFS) and overall survival (OS); the secondary endpoint includes objective response rate (ORR), disease control rate (DCR) and safety

ELIGIBILITY:
Inclusion Criteria:

* Age: ≥18 years old
* Gender: no limitation
* Diagnosed as primary hepatocellular carcinoma histologically or clinically
* Imaging data within 31 days at enrollment and at least one measurable lesion (according to mRECIST criteria) is available
* Patients only received treatment with HepaSphere combined with hepatocellular arterial infusion chemotherapy (HAIC) or HAIC alone during the observation period
* Child-Pugh: A-B
* ECOG: 0-2.

Exclusion Criteria:

* Other cancer diseases are co-existed
* Drug-eluting beads from other manufacturers were used during DEB-TACE
* DEB-TACE combined with HAIC or HAIC alone was used as postoperative adjuvant therapy
* Pre- or post-surgery relevant examination results were unavailable
* Imaging information for effectiveness evaluation was unavailable
* Follow-up failure due to patient information errors, loss, refusal, etc

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all of patients were diagnosed as HCC. Some of them may received the treatment before enrollment. They only received HepaSphere plus HAIC or HAIC alone as the interventional therapy during this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-Free Survival (PFS) | Up to 3 year
  Progression-free survival is defined as the time from the start of treatment DEB-TACE plus HAIC or HAIC until the first documentation of disease progression or death due to any cause, whichever occurs first
Overall Survival (OS) | Up to 3 year
  Overall survival is defined as the time from the start of treatment with DEB-TACE plus HAIC or HAIC until death due to any cause

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to 3 year
  The ORR is defined as the proportion of subjects with confirmed CR or confirmed PR, based on RECIST Version 1.1
Duration of Response (DoR) | Up to 3 years
  Duration of response is defined as the duration from the first documentation of objective response to the first documented disease progression or death due to any cause, whichever occurs first

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No